CLINICAL TRIAL: NCT05893745
Title: Effectiveness of Dermoneuromodulation Techniques in Patients With Non-specific Chronic Neck Pain: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/07EGY10000
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Cervical Pain; Cervical
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Supervised Exercise Program
  Interventions: Other: Supervised Exercise Program
- Study Group (Experimental): Combination of Exercise and Dermoneuromodulation Techniques
  Interventions: Other: Supervised Exercise Program plus Dermoneuromodulation Techniques

INTERVENTIONS:
Other: Supervised Exercise Program — Participants in the control group will receive a supervised exercise program that consists of three weekly sessions in addition to home exercises, over the course of four weeks. This program will include stabilization, flexing, extension, and rotation exercises for the cervical region and self-mobilization targeting the deep neck muscles. Participants will be instructed to perform the exercises at home three times a week in a manner that did not cause pain.
  Arms: Control Group
Other: Supervised Exercise Program plus Dermoneuromodulation Techniques — Participants in the study group will receive the same supervised exercise program as the control group, with home exercises, in addition to two dermoneuromodulation techniques for the Dorsal Cutaneous Nerve (C3-T1), which are the skin stretch technique and kitten technique. Patients in this group will receive 3 sessions/week for a total of 4 weeks.
  Arms: Study Group

SUMMARY:
PURPOSE: The purpose of the present study is to investigate the benefit of applying dermoneuromodulation techniques in patients with non-specific chronic neck pain.

BACKGROUND: Chronic neck pain is one of the most commonly reported musculoskeletal pathologies in the general population. It has an immense impact on the physical, social, and psychological aspects and quality of life of the individual and society as a whole. Dermoneuromodulation(DNM) is recently popularising touch based pain relieving approach which is a gentle, structured method of interacting with patient's nervous system to help them resolve pain, regain function, and feel better. It was developed by Diane Jacobs, a Canadian physiotherapist specialised in pain science and the treatment of painful conditions. During her 40 years of practice, Jacobs was interested in Ronald Melzack, who developed the original Gate Control theory of pain along with Patrick Wall, and who later developed the NeuroMatrix model of pain. In 2007, Jacobs made a cadaver study that defined how peripheral cutaneous nerves divide into rami, which spread outward into the underside of skin. This work inspired her to develop a new conceptual approach to manual therapy for patients with pain.

HYPOTHESES We hypothesize that there will be no effect of dermoneuromodulation techniques on clinical outcomes of patients with non-specific chronic neck pain.

RESEARCH QUESTION: Is there a statistically significant effect of dermoneuromodulation techniques on clinical outcomes of patients with non-specific chronic neck pain?

ELIGIBILITY:
Inclusion Criteria:

* Recurrent history of non-specific chronic neck pain (NSCNP) of not less than 3 months duration.
* Pain level greater than or equal to 5/10 on the Numeric Pain Rating Scale (NPRS).
* Age between 25 to 40 years.
* Both male and female participants.
* Diagnosis of non-specific chronic neck pain confirmed by a licensed physiotherapist or physician using a combination of the following criteria:
* Absence of specific pathologies or conditions causing neck pain (e.g., disc prolapse, tumor of the cervical spine, whiplash injury, cervical fractures, or cervicogenic headache) as assessed by clinical examination and medical history.
* Presence of at least three of the following signs and symptoms:

  1. Restricted cervical range of motion.
  2. Pain provoked or increased with neck movement or sustained neck postures.
  3. Palpable muscle tension or tenderness in the neck or upper back region.
  4. Referred pain or symptoms to the shoulders, upper back, or arms.
* Neck pain not attributed to a specific cause after careful evaluation, including imaging studies (e.g., X-ray, MRI, or CT scan) if deemed necessary by the clinician.

Exclusion Criteria:

* Serious pathology such as specific neck pain due to disc prolapse, tumor of the cervical spine, whiplash injury, cervical fractures, or cervicogenic headache.
* Any neurological signs consistent with nerve root compression.
* Prior surgery in the cervical region.
* Inability to comply with the exercise program or attend scheduled sessions.
* Contraindications to dermoneuromodulation techniques, such as active skin infections or severe inflammatory skin conditions.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Numeric Pain Rating Scale (NPRS) | Baseline, 2 weeks post-treatment, 4 weeks post-treatment, and 3 months post-treatment.
  The NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) to measure the intensity of pain.
Changes in Neck Disability Index (NDI) | Baseline, 2 weeks post-treatment, 4 weeks post-treatment, and 3 months post-treatment.
  The NDI is a 10-item questionnaire used to measure functional disability related to neck pain. Each item is scored from 0 to 5, with a total possible score of 50. Higher scores indicate greater disability.

SECONDARY OUTCOMES:
Chnages in Pressure Pain Threshold (PPT) | Baseline, 2 weeks post-treatment, 4 weeks post-treatment, and 3 months post-treatment.
  The PPT is a measure of the minimum amount of pressure applied to a specific location that elicits pain. It is assessed using a handheld pressure algometer.
Changes in cervical range of motion | Baseline, 2 weeks post-treatment, 4 weeks post-treatment, and 3 months post-treatment.
  The CROM is a measure of the movement in degrees around each axis (flexion, extension, lateral flexion, and rotation) of the cervical spine. It is assessed using a CROM device.
Changes in Fear-Avoidance Beliefs Questionnaire (FABQ) | Baseline, 2 weeks post-treatment, 4 weeks post-treatment, and 3 months post-treatment.
  The FABQ is a 16-item questionnaire used to assess fear-avoidance beliefs related to physical activity and work in patients with musculoskeletal pain. The score ranges from 0 to 96, with higher scores indicating greater fear-avoidance beliefs.
Changes in Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 2 weeks post-treatment, 4 weeks post-treatment, and 3 months post-treatment.
  The PSEQ is a 10-item questionnaire used to assess the confidence of individuals with chronic pain in performing activities while in pain. The score ranges from 0 to 60, with higher scores indicating greater pain self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The researchers of this study are committed to promoting open science and collaboration among researchers. As part of this commitment, we will share de-identified individual participant data (IPD) with other qualified researchers, upon request and in accordance with applicable regulations and ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD will be available for sharing with other researchers starting six months after the publication of the primary study results and will remain accessible for a period of five years.
Access Criteria: mohamed.elmeligie@acu.edu.eg